CLINICAL TRIAL: NCT07369427
Title: Magnetic Tracking and Electrocardiography-Guided Tip Confirmation System for Placement of Peripherally Inserted Central Catheters
Brief Title: Magnetic Tracking and ECG-Guided Tip Confirmation System for PICCs
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zeyin Hu, Project Researcher, Sun Yat-sen University
Other Study IDs: SunYat-senU6
Record Dates: First submitted 2025-09-27; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: Peripherally Inserted Central Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer patients who undergo PICC placement (Caprini score ≥5)
  Interventions: Other: Sherlock 3CG Tip Confirmation System

INTERVENTIONS:
Other: Sherlock 3CG Tip Confirmation System — Sherlock 3CG Tip Confirmation System: An integrated system combining magnetic navigation tracking and ECG guidance. It dynamically confirms the tip's position relative to the target anatomical location (e.g., superior vena cava-right atrial junction) by real-time tracking of the catheter tip's spatial position via magnetic navigation and synchronously monitoring ECG signals (e.g., P-wave changes).
  Traditional ECG-Guided Tip Positioning Technology: Relying solely on ECG monitoring for guidance, it assists in determining the tip position via characteristic waveform changes in intracardiac ECG signals (e.g., changes in P-wave amplitude) derived from the catheter tip electrode as the tip approaches the target location, serving as a conventional positioning method.

SUMMARY:
This prospective study enrolled cancer patients who underwent peripherally inserted central catheter (PICC) placement at a tertiary care oncology hospital in Guangzhou between January 1st and May 30th, 2026. Data on catheterization outcomes and complications were collected to compare two tip positioning techniques: electromagnetic navigation tip positioning and traditional electrocardiogram (ECG)-guided positioning. The outcomes assessed included first-attempt catheterization success rate, tip positioning accuracy, catheterization procedure time, post-procedural catheter adjustment time, and the incidence of complications (thrombosis, infection, and catheter dysfunction) within 4 weeks post-catheterization.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients receiving PICC placement
* High risk of PICC-related thrombosis(Evaluated by Caprini score ≥ 5)
* Agree to receive PICC maintenance at the research hospital;
* Sign the informed consent form

Exclusion Criteria:

* PICC placed in the lower limb
* Estimated survival time less than one month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who receiving PICC placement
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
one time catheterization rate | data will be collected on Day 1

SECONDARY OUTCOMES:
time for catheter tip positioning during catheterization | on Day 1
time for catheter tip adjustment after catheterization | on Day 1
rate of correct catheter tip positioning | on Day 1
rate of PICC-related complications | within 4 weeks after catheterization

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-08-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT07369427/ICF_000.pdf